CLINICAL TRIAL: NCT01144767
Title: Computer-Based Physical Activity Advice for Ethnic Minority Aging Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Northeastern University (Other)
Responsible Party: Principal Investigator, Abby C King, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SU-04262010-5762; 10894
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Communication; Health Behavior; Sedentary Lifestyle
MeSH Terms: conditions — Communication; Health Behavior; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer-generated advisor (Experimental): Participants receive sessions with a computer-generated adviser who will provide tailored advice and encouragement to engage in physical activity.
  Interventions: Behavioral: Computer-generated advisor
- Comparison control condition (Active Comparator): Participants will receive live, group sessions on health topics unrelated to physical activity.
  Interventions: Behavioral: Comparison control condition

INTERVENTIONS:
Behavioral: Computer-generated advisor — Weekly sessions with a computer generated advisor who offers advice, feedback and guidance on physical activity
  Arms: Computer-generated advisor
Behavioral: Comparison control condition — Weekly/biweekly sessions with a group facilitator to receive health education and information.
  Arms: Comparison control condition

SUMMARY:
Despite the recognized health benefits of a physically active lifestyle, mid-life and older low-income and ethnic minority adults, including Hispanic Americans, are among the least active and understudied groups in the U.S. This research aims to develop and evaluate a bi-lingual physical activity promotion program, applying easy to use state-of-the-art computer technology, which is tailored to the preferences and needs of mid-life and older Latino adults. Such computer-based programs represent a potentially low-cost means for reaching the large proportion of low-income and ethnic minority Americans who are under-active.

DETAILED DESCRIPTION:
During Phase 1 of this study, the computer program will be adapted to better help Latino older adults to increase physical activity levels. Researchers will conduct focus groups and/or individual interviews to obtain participants feedback used to tailor the program to be appropriate for this population.

During Phase 2, the computer-generated adviser program will be tested to see if it is effective in promoting an increase in physical activity (primarily walking) levels among Latino older adults.

Participants will be randomly assigned to use the computer-generated adviser or to the wait list control group. Participants in the embodied conversational agent (computer-generated adviser) group receive an initial session with a staff health educator to review the expectations and content of this walking program. They will learn how to log onto the computer and interact with the computer adviser using a touch-screen. Participants will interact with the computer adviser at least 3 times per week to report past physical activity (primarily walking) completed, review obstacles (or barriers) to walking, and to set future walking goals. They are also asked to wear a pedometer.

Participants assigned to the wait list will receive an initial session with a staff health educator to review the expectations and content of this program. They will attend a monthly interactive class-based group session lead by a health educator that will cover health-related topics relevant for the older adult such as nutrition, stress management, and brain health. At the end of their involvement with this group they can decide if they want to use the computer adviser program.

Participants of both groups complete physical activity and computer-related questionnaires at the beginning (at 2 months) and at the end of the study (4 months).

ELIGIBILITY:
Inclusion Criteria:1. Spanish or English-speaking Latino men or women 2. Greater than or equal to 55 years of age 3. No plans to move within the next year 4. Inactive (have not engaged in moderate-intensity or more vigorous physical activity, > 3 days per week for at least 20 min per day) within last 6-months 5. Able to participate in study intervention and assessments at the community-based location 6. Willing to be randomly assigned to either study arm (Year 02) Exclusion Criteria:1. Any medical condition or disorder that would limit participation in moderate intensity physical activity (such as sustained walking), including life-threatening disorders, myocardial ischemia, and major functional disabilities in the orthopedic area 2. Not stable on their medications, including hormone replacement therapy, for 3 months 3. Severe depressive symptomatology (score > 16 on the 18-item Spanish version of the Center for Epidemiologic Studies Depression Scale [CES-D]); English version used when indicated 4. Gross levels of dementia (score< 23 on the Folstein Mini-Mental State Exam) 5. Inability to complete a face-to-face training session with the embodied conversational agent (ECA) program

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Community Healthy Activities Model Program for Seniors (CHAMPS) Questionnaire | 4 months
  self-report questionnaire to assess frequency and quantity of physical activity
steps per day measured by accelerometry | 4 months
  objective measure of physical activity collected by accelerometer monitor

SECONDARY OUTCOMES:
physical activity self-efficacy | 4 months
  self-report questionnaire of perceived confidence to engage in physical activity under a variety of circumstances
physical activity decisional balance | 4 months
  self-report questionnaire of perceived pros and cons of engaging in physical activity
Computer Attitude Scale | 4 months
  self-report questionnaire of perceived confidence and anxiety around computers and technology
Working Alliance Inventory | 4 months
  self-report questionnaire of perceptions and attitudes about the working relationship with the advisor

CONTACTS AND LOCATIONS:
Overall Officials: Abby C King, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] King AC, Bickmore TW, Campero MI, Pruitt LA, Yin JL. Employing virtual advisors in preventive care for underserved communities: results from the COMPASS study. J Health Commun. 2013;18(12):1449-64. doi: 10.1080/10810730.2013.798374. Epub 2013 Aug 13. PMID 23941610